CLINICAL TRIAL: NCT01246427
Title: Placebo-controlled Evaluation of the Homeopathic Drug BRN01 for the Treatment of Hot Flashes in Women With Non Metastatic Breast Cancer Treated by Adjuvant Hormonal Therapy
Brief Title: Evaluation of Homeopathic Treatment for Hot Flashes in Non Metastatic Breast Cancer
Acronym: HBC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: BOIRON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBC; ET2008-048
Record Dates: First submitted 2010-11-16; First posted 2010-11-23 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Adjuvant hormonal therapy; Homeopathic treatment; Hot flashes; Quality of life; Hot flash score
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BRN01 (Experimental): A 2 to 4 weeks run-in period is planned, during which all patients receive single blinded "hot flash evaluation treatment" which is actually a placebo (2 tablets every morning and every evening during 2 to 4 weeks). At the end of this period, the hot flash score is calculated. If the score is ≥10, the patient can be randomized to one of the 2 arms:
  * Experimental: BRN01
  * Placebo Comparator: Placebo
  Interventions: Drug: BRN01
- Placebo (Placebo Comparator): A 2 to 4 weeks run-in period is planned, during which all patients receive single blinded "hot flash evaluation treatment" which is actually a placebo (2 tablets every morning and every evening during 2 to 4 weeks). At the end of this period, the hot flash score is calculated. If the score is ≥10, the patient can be randomized to one of the 2 arms:
  * Experimental: BRN01
  * Placebo Comparator: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRN01 — 2 tablets every morning and every evening during 8 to 10 weeks. Each patient will receive 1 set of 5 treatment boxes (60 tablets/box).
  Arms: BRN01
Drug: Placebo — 2 tablets every morning and every evening during 8 to 10 weeks. Each patient will receive 1 set of 5 treatment boxes (60 tablets/box).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of a homeopathic treatment (BRN01) in reducing hot flash scores after 4 weeks of treatment.

DETAILED DESCRIPTION:
Chemotherapy is used as an adjuvant treatment for breast cancer, like hormone therapy in patients with hormone-sensitive breast cancer or immunotherapy in those with Human Epidermal growth factor Receptor 2 (HER2)-overexpressing cancer.

These adjuvant treatments reduce the risk of recurrence and metastasis. The side effects of hormone therapy are known and depend on the therapeutic strategy and the drugs used. The side effects of Tamoxifen are similar to menopausal symptoms: hot flashes (half of the female population), vaginal dryness or leukorrhea, nausea, irregular menstruation, benign ovarian cyst and, less frequently, weight gain. Aromatase inhibitors have the same side effects, though with lesser frequency and intensity. The incidence rate of hot flashes after adjuvant treatment in menopausal women with localized breast cancer is 60 to 65 %, and these reactions are very severe in one third of these women. Despite this fact, the management of hot flashes is not systematic and there is currently no therapeutic strategy with proven efficiency. BRN01 (Boiron laboratory) is a homeopathic remedy whose active ingredient is already present in other homeopathic drugs indicated for the management of menopausal hot flashes. BRN01 could reduce the intensity of the reaction in women with breast cancer receiving adjuvant hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patient aged ≥ 18 years
* Women with histologically proven non metastatic breast cancer
* ECOG PS ≤ 1
* Patient receiving adjuvant hormonal therapy for at least 1 month (aromatase inhibitor or Tamoxifen ± ovarian function suppression (Luteinizing Hormone Releasing Hormone agonist (LH-RH agonist), ovariectomy...))
* Patient complaining of hot flashes with moderate to severe intensity, affecting quality of life, for at least 1 month before inclusion
* Patient agreement not to start another hot flash treatment during the study (allopathic treatment, E vitamin, dietary supplement, phytotherapy, acupuncture...)
* Patient able to understand, read and write French
* Mandatory affiliation with a health insurance system
* Signed, written informed consent

Exclusion Criteria:

* Ongoing chemotherapy or radiotherapy, or treatment planned to begin during the study
* Patient with a condition known to induce hot flashes such as hyperthyroidism, diabetes, adrenal tumor, enteric carcinoid tumor, mastocytosis...
* Patient with severe renal failure, severe hepatic failure, or cardiovascular disease
* Patient with one of the following contraindications:

  * known hypersensitivity to one of the components of the study drug
  * galactose, fructose intolerance
  * Lapp lactase deficiency, isomaltase invertase deficiency
  * Glucose or galactose malabsorption syndrome
* Follow up impossible because of social, familial, geographical or psychological reasons
* Patient suspected of poor compliance with protocol or treatment
* Participation in another biomedical research trial in the same indication, or administration of an experimental drug in the same indication in the 30 days before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-01; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of BRN01 efficacy in reducing hot flash score after 4 weeks of treatment | The patients are instructed to record the number and intensity of hot flashes in a self-evaluation booklet every day during the 2nd week of the first period (run-in period) and during the 4th week of the second period (placebo or BRN01).
  The hot flash score is equal to: (number of hot flashes/day) x (mean intensity/day).
  Treatment efficiency scores will be calculated as follows: (hot flash score on the 4th week of the second period)-(hot flash score on the 2nd week of the first period).
  Then efficiency scores will be compared between the 2 arms (placebo versus BRN01).

SECONDARY OUTCOMES:
Evaluation of BRN01 efficacy in reducing the hot flash score after 8 weeks of treatment | The patients are instructed to record the number and intensity of hot flashes in a self-evaluation booklet every day during the 2nd week of the first period (run-in period) and during the 8th week of the second period (placebo or BRN01).
  Treatment efficacy scores will be calculated as follows: (hot flash score on the 8th week of the second period)-(hot flash score on the 2nd week of the first period).
  Then efficiency scores will be compared between the 2 arms (placebo versus BRN01).
Evaluation of the mean daily intensity of hot flashes during the run-in period and on the 4th and 8th weeks of treatment in both arms. | The patients are instructed to record the intensity of hot flashes in a self-evaluation booklet, daily, during the 2nd week of the first period (run-in period), and during the 4th and 8th weeks of the second period (placebo or BRN01).
Evaluation of the mean daily frequency of hot flashes during the run-in period and on the 4th and 8th weeks of treatment in both arms. | The patients are instructed to record the number of hot flashes in a self-evaluation booklet, daily, during the 2nd week of the first period (run-in period), and during the 4th and 8th weeks of the second period (placebo or BRN01).
Evaluation of quality of life in both arms | The patients are instructed to complete quality of life items on the 7th day of each evaluation period (2nd week of the run-in period, 4th and 8th weeks of the second period)
Evaluation of patient satisfaction with the treatment and with the management of hot flashes. | The patients are instructed to record all new hot flash treatments started, as well as their satisfaction with their management, on the 7th day of each evaluation period (2nd week of the run-in period, 4th and 8th weeks of the second period).
Evaluation of treatment tolerance | Side effects are registered by the oncologist at each visit (planned during the 3rd week or the 4th week of the run-in period and during the 9th week or the 10th week of the second period)
Evaluation of patient compliance | The number of remaining tablets will be counted at each visit (planned during the 3rd week or the 4th week of the run-in period and during the 9th week or the 10th week of the second period)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Etienne Heudel, MD, Principal Investigator — Centre Leon Berard, France
Locations (9):
- France (9):
  - Centre Hospitalier de Chambery, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Centre Hospitalier de Montelimar, Montélimar
  - Centre Hospitalier d'Annecy, Pringy
  - Centre Hospitalier de Roanne, Roanne
  - Clinique Armoricaine de radiologie, Saint-Brieuc
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Hospitalier de Valence, Valence

REFERENCES:
- [Background] Remontet L, Esteve J, Bouvier AM, Grosclaude P, Launoy G, Menegoz F, Exbrayat C, Tretare B, Carli PM, Guizard AV, Troussard X, Bercelli P, Colonna M, Halna JM, Hedelin G, Mace-Lesec'h J, Peng J, Buemi A, Velten M, Jougla E, Arveux P, Le Bodic L, Michel E, Sauvage M, Schvartz C, Faivre J. Cancer incidence and mortality in France over the period 1978-2000. Rev Epidemiol Sante Publique. 2003 Feb;51(1 Pt 1):3-30. PMID 12684578
- [Background] Menegoz F, Black RJ, Arveux P, Magne V, Ferlay J, Buemi A, Carli PM, Chapelain G, Faivre J, Gignoux M, Grosclaude P, Mace-Lesec'h J, Raverdy N, Schaffer P. Cancer incidence and mortality in France in 1975-95. Eur J Cancer Prev. 1997 Oct;6(5):442-66. doi: 10.1097/00008469-199710000-00005. PMID 9466116
- [Background] Coleman MP. Trends in breast cancer incidence, survival, and mortality. Lancet. 2000 Aug 12;356(9229):590-1; author reply 593. doi: 10.1016/S0140-6736(00)02593-9. No abstract available. PMID 10950250
- [Background] Breast International Group (BIG) 1-98 Collaborative Group; Thurlimann B, Keshaviah A, Coates AS, Mouridsen H, Mauriac L, Forbes JF, Paridaens R, Castiglione-Gertsch M, Gelber RD, Rabaglio M, Smith I, Wardley A, Price KN, Goldhirsch A. A comparison of letrozole and tamoxifen in postmenopausal women with early breast cancer. N Engl J Med. 2005 Dec 29;353(26):2747-57. doi: 10.1056/NEJMoa052258. PMID 16382061
- [Background] Finck G, Barton DL, Loprinzi CL, Quella SK, Sloan JA. Definitions of hot flashes in breast cancer survivors. J Pain Symptom Manage. 1998 Nov;16(5):327-33. doi: 10.1016/s0885-3924(98)00090-6. PMID 9846028
- [Background] Stearns V, Ullmer L, Lopez JF, Smith Y, Isaacs C, Hayes D. Hot flushes. Lancet. 2002 Dec 7;360(9348):1851-61. doi: 10.1016/s0140-6736(02)11774-0. PMID 12480376
- [Background] Couzi RJ, Helzlsouer KJ, Fetting JH. Prevalence of menopausal symptoms among women with a history of breast cancer and attitudes toward estrogen replacement therapy. J Clin Oncol. 1995 Nov;13(11):2737-44. doi: 10.1200/JCO.1995.13.11.2737. PMID 7595732
- [Background] Fellowes D, Fallowfield LJ, Saunders CM, Houghton J. Tolerability of hormone therapies for breast cancer: how informative are documented symptom profiles in medical notes for 'well-tolerated' treatments? Breast Cancer Res Treat. 2001 Mar;66(1):73-81. doi: 10.1023/a:1010684903199. PMID 11368413
- [Background] Lower EE, Blau R, Gazder P, Tummala R. The risk of premature menopause induced by chemotherapy for early breast cancer. J Womens Health Gend Based Med. 1999 Sep;8(7):949-54. doi: 10.1089/jwh.1.1999.8.949. PMID 10534297
- [Background] McPhail G, Smith LN. Acute menopause symptoms during adjuvant systemic treatment for breast cancer: a case-control study. Cancer Nurs. 2000 Dec;23(6):430-43. doi: 10.1097/00002820-200012000-00005. PMID 11128122
- [Background] Loprinzi CL, Zahasky KM, Sloan JA, Novotny PJ, Quella SK. Tamoxifen-induced hot flashes. Clin Breast Cancer. 2000 Apr;1(1):52-6. doi: 10.3816/cbc.2000.n.004. PMID 11899390
- [Background] Love RR, Cameron L, Connell BL, Leventhal H. Symptoms associated with tamoxifen treatment in postmenopausal women. Arch Intern Med. 1991 Sep;151(9):1842-7. PMID 1888251
- [Background] Linde K, Clausius N, Ramirez G, Melchart D, Eitel F, Hedges LV, Jonas WB. Are the clinical effects of homeopathy placebo effects? A meta-analysis of placebo-controlled trials. Lancet. 1997 Sep 20;350(9081):834-43. doi: 10.1016/s0140-6736(97)02293-9. PMID 9310601
- [Background] Jonas WB, Kaptchuk TJ, Linde K. A critical overview of homeopathy. Ann Intern Med. 2003 Mar 4;138(5):393-9. doi: 10.7326/0003-4819-138-5-200303040-00009. PMID 12614092
- [Background] Cucherat M, Haugh MC, Gooch M, Boissel JP. Evidence of clinical efficacy of homeopathy. A meta-analysis of clinical trials. HMRAG. Homeopathic Medicines Research Advisory Group. Eur J Clin Pharmacol. 2000 Apr;56(1):27-33. doi: 10.1007/s002280050716. PMID 10853874
- [Background] Jonas WB. Researching alternative medicine. Nat Med. 1997 Aug;3(8):824-7. doi: 10.1038/nm0897-824. No abstract available. PMID 9256264
- [Background] Guyatt GH, Sackett DL, Cook DJ. Users' guides to the medical literature. II. How to use an article about therapy or prevention. A. Are the results of the study valid? Evidence-Based Medicine Working Group. JAMA. 1993 Dec 1;270(21):2598-601. doi: 10.1001/jama.270.21.2598. No abstract available. PMID 8230645
- [Background] Grol R, Grimshaw J. Evidence-based implementation of evidence-based medicine. Jt Comm J Qual Improv. 1999 Oct;25(10):503-13. doi: 10.1016/s1070-3241(16)30464-3. PMID 10522231
- [Background] Barnes J, Ernst E. Complementary medicine. Br J Gen Pract. 1997 May;47(418):329. No abstract available. PMID 9219418
- [Background] Clover A, Ratsey D. Homeopathic treatment of hot flushes: a pilot study. Homeopathy. 2002 Apr;91(2):75-9. doi: 10.1054/homp.2002.0004. PMID 12371460
- [Background] Thompson EA, Reilly D. The homeopathic approach to the treatment of symptoms of oestrogen withdrawal in breast cancer patients. A prospective observational study. Homeopathy. 2003 Jul;92(3):131-4. doi: 10.1016/s1475-4916(03)00035-3. PMID 12884894
- [Background] Thompson EA, Montgomery A, Douglas D, Reilly D. A pilot, randomized, double-blinded, placebo-controlled trial of individualized homeopathy for symptoms of estrogen withdrawal in breast-cancer survivors. J Altern Complement Med. 2005 Feb;11(1):13-20. doi: 10.1089/acm.2005.11.13. PMID 15750359
- [Background] Relton C, Weatherley-Jones E. Homeopathy service in a National Health Service community menopause clinic: audit of clinical outcomes. J Br Menopause Soc. 2005 Jun;11(2):72-3. doi: 10.1258/136218005775544516. PMID 15970019
- [Background] Bordet MF, Colas A, Marijnen P, Masson J, Trichard M. Treating hot flushes in menopausal women with homeopathic treatment--results of an observational study. Homeopathy. 2008 Jan;97(1):10-5. doi: 10.1016/j.homp.2007.11.005. PMID 18194760
- [Background] Sloan JA, Loprinzi CL, Novotny PJ, Barton DL, Lavasseur BI, Windschitl H. Methodologic lessons learned from hot flash studies. J Clin Oncol. 2001 Dec 1;19(23):4280-90. doi: 10.1200/JCO.2001.19.23.4280. PMID 11731510
- [Derived] Heudel PE, Van Praagh-Doreau I, Duvert B, Cauvin I, Hardy-Bessard AC, Jacquin JP, Stefani L, Vincent L, Dramais D, Guastalla JP, Blanc E, Belleville A, Lavergne E, Perol D. Does a homeopathic medicine reduce hot flushes induced by adjuvant endocrine therapy in localized breast cancer patients? A multicenter randomized placebo-controlled phase III trial. Support Care Cancer. 2019 May;27(5):1879-1889. doi: 10.1007/s00520-018-4449-x. Epub 2018 Sep 7. PMID 30194492